CLINICAL TRIAL: NCT04240574
Title: Evaluation of Micro Water Jet Technology and the Progression of Wound Healing: A Prospective Cohort Evaluating the Efficacy of Micro Water Jet Technology in the Debridement and Healing of Chronic Lower Extremity Ulcers
Brief Title: Debritom - Micro Water Jet Technology and Wound Healing
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Due to pandemic we were not able to recruit patients for this study
Sponsor: Stephanie Wu (Other)
Responsible Party: Sponsor-Investigator, Stephanie Wu, Principal Investigator, Rosalind Franklin University of Medicine and Science
Organization: Rosalind Franklin University of Medicine and Science (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MDX-DEB-001
Record Dates: First submitted 2020-01-06; First posted 2020-01-27 (Actual); Results first posted 2023-03-27 (Actual); Last update posted 2023-03-27 (Actual); Status verified 2023-03

CONDITIONS: Diabetic Foot Ulcer; Non-healing Wound; Non-Healing Ulcer of Skin; Venous Leg Ulcer; Venous Ulcer
MeSH Terms: conditions — Diabetic Foot; Varicose Ulcer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (1):
- Micro Water Jet Technology (Debritom) (Other): Debritom is a hydrosurgery device that utilizes micro water jet technology that has been designed to debride acute and chronic wounds precisely and in a tissue-preserving manner.
  All subject will get the Debritom.
  Interventions: Device: Debritom

INTERVENTIONS:
Device: Debritom — hydrosurgery device that utilizes micro water jet technology that has been designed to debride acute and chronic wounds precisely and in a tissue-preserving manner.

SUMMARY:
This study will investigate the clinical efficacy of micro water jet technology in the debridement and healing of chronic lower extremity ulcers.

DETAILED DESCRIPTION:
This is a prospective cohort, single-center, open-label study in subjects with chronic lower extremity wounds. The study will enroll up to 20 subjects. Subjects will undergo screening evaluations to determine eligibility to enroll in the study. All study subjects will receive micro water jet technology debridement as opposed to other debridement methods as part of their wound care treatment. The other aspects of subjects wound care protocol will remain unchanged. In the case of bilateral limb ulcers, or multiple ulcers, subjects will have the option to receive micro water jet debridement on one or all of the ulcers.

ELIGIBILITY:
Inclusion Criteria:

* Male or female age 18 or older
* The ability and willingness to provide Informed consent
* Presence of a chronic lower extremity ulcer
* Chronic ulcer is defined as that greater than 4 weeks in duration.
* Subject's informed consent for participation prior to proceeding with micro water jet technology debridement
* Patient's ulcer cannot exhibit any gross clinical signs of infection.
* Patient is willing to participate in all procedures and follow up evaluations necessary to complete the study.
* Patient willing and able to comply with having micro water jet technology debridement potentially weekly or biweekly as part of their wound care treatment plan for up to 20 weeks.

Exclusion Criteria:

* Patients with active wound infection, or untreated osteomyelitis
* Patients with dementia, or impaired cognitive function
* Patients who are unable or unwilling to participate in all procedures and follow up evaluations
* Patient has Active Charcot foot
* Patient with malignant wounds

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2020-01-24 (Actual); Primary Completion 2021-08-06 (Actual); Study Completion 2021-08-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Rosalind Franklin University Health Clinics, North Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
Will not share

RESULTS

PARTICIPANT FLOW:
Groups:
- Participants: Up to 20 participants may be recruited.
Period: Overall Study
Arm/Group | Participants
Started | 2 (Due to the pandemic we were only able to recruit 2 participants. Study was terminated early due to the pandemic.)
Completed | 2 (Due to the pandemic we were only able to recruit 2 participants. Study was terminated early due to the pandemic.)
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Unable to complete the study due to national pandemic. We were only able to have two participants.
Groups:
- Study Treatments: All study subjects will receive micro water jet technology debridement as opposed to traditional debridement using instruments or other means of debridement. Other aspects of subjects wound care protocol will remain unchanged.
Arm/Group | Study Treatments
Number analyzed (Participants) | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 2
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  United States | 2

OUTCOME MEASURES:

1. Primary Outcome: Size of Ulcers
Description: The extent and size of ulcers (summation of the products of the long x short axis for all ulcers measured in centimeters squared, plus ulcer depth) will be evaluated and photographs of ulcers taken during screening and on all clinic visits up to 20 weeks or when the ulcer is healed, whichever is sooner.
Time Frame: Up to 20 weeks or when the ulcer is healed, whichever is sooner.
Population: Data not collected.
Groups:
- Size of Ulcers: The extent and size of ulcers (summation of the products of the long x short axis for all ulcers measured in centimeters squared, plus ulcer depth) will be evaluated and photographs of ulcers taken during screening and on all clinic visits
Arm/Group | Size of Ulcers
Number analyzed (Participants) | 0

2. Primary Outcome: Leg Rest Pain Score
Description: Leg rest pain score - visual analogue scale (VAS) graded from 0 (pain free) to Grade 10 (maximum pain) during screening and on all clinic visits up to 20 weeks, or when the ulcer is healed, whichever is sooner.
Time Frame: up to 20 weeks, or when the ulcer is healed, whichever is sooner
Population: Data not collected.
Groups:
- Pain Score: Leg rest pain score - visual analogue scale (VAS) graded from 0 (pain free) to Grade 10 (maximum pain) during screening and on all clinic visits up to 20 weeks, or when the ulcer is healed, whichever is sooner.
Arm/Group | Pain Score
Number analyzed (Participants) | 0

3. Primary Outcome: Pain During Debridement Score
Description: Pain during Debridement score - VAS graded from 0 (pain free) to Grade 10 (maximum pain) during on all clinical visits when debridement is performed for up to 20 weeks, sooner pending wound healing.
Time Frame: up to 20 weeks, sooner pending wound healing.
Population: Data not collected.
Groups:
- Pain During Debridement Score: VAS graded from 0 (pain free) to Grade 10 (maximum pain) during on all clinical visits when debridement is performed
Arm/Group | Pain During Debridement Score
Number analyzed (Participants) | 0

4. Primary Outcome: Subjects Feedback
Description: Subjects feedback regarding their debridement experience with micro water jet technology will be collected on all clinical visits when debridement is performed.
Time Frame: At end of their study participation
Population: Data not collected.
Groups:
- Subject Feedback: Subjects feedback regarding their debridement experience with micro water jet technology will be collected on all clinical visits when debridement is performed.
Arm/Group | Subject Feedback
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Six months.
Groups:
- All Participants: All participants, which was only two for this study due study terminating due to the pandemic.
Arm/Group | All Participants
All-Cause Mortality (participants affected / at risk) | 0/2
Serious Adverse Events (participants affected / at risk) | 0/2
Other Adverse Events (participants affected / at risk) | 0/2

LIMITATIONS AND CAVEATS:
Early termination of study due to pandemic. The study was not able to be completed.

The early termination lead to only two subjects taking part of the study.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-09-30): https://cdn.clinicaltrials.gov/large-docs/74/NCT04240574/Prot_SAP_002.pdf
  • Informed Consent Form (2019-09-30): https://cdn.clinicaltrials.gov/large-docs/74/NCT04240574/ICF_001.pdf